CLINICAL TRIAL: NCT00944307
Title: Effect of Antacids on the Pharmacokinetics of Raltegravir in Healthy Volunteers
Brief Title: Effect of Antacids on the Pharmacokinetics of Raltegravir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 09-0475
Record Dates: First submitted 2009-07-20; First posted 2009-07-23 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: HIV Infections
Keywords: HIV; antiretroviral; drug interaction; human immunodeficiency virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; Antacids; aluminum hydroxide, magnesium hydroxide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- raltegravir alone (Active Comparator): Subjects will receive a single dose of 400 mg raltegravir orally
  Interventions: Drug: raltegravir
- raltegravir plus antacid (Experimental): Subjects will receive a single dose of 400mg raltegravir orally simultaneously with an antacid
  Interventions: Drug: raltegravir; Drug: antacid

INTERVENTIONS:
Drug: raltegravir — raltegravir 400mg orally once
  Other Names: Isentress
Drug: antacid — aluminum, magnesium, simethicone-containing antacid 30mL orally once
  Other Names: Isentress, Maalox Plus Extra Strength
  Arms: raltegravir plus antacid

SUMMARY:
The purpose of this study is to test whether there is a drug interaction between raltegravir (a medicine used to treat the human immunodeficiency virus or HIV) and antacids.

DETAILED DESCRIPTION:
This study will determine if an interaction occurs between the HIV medicine raltegravir and an antacid. A prior study found an interaction with another medicine like raltegravir called elvitegravir and an antacid. The elvitegravir levels were reduced by half. The same interaction may occur with raltegravir and an antacid based on the structure of this medicine and how it works. When the levels of HIV medications are reduced, people with HIV can "fail" their treatment. The virus can multiply when the drug levels are too low and the medications can stop working. We need to be sure that antacids will not cause this problem with raltegravir.

ELIGIBILITY:
Inclusion Criteria:

* Absence of HIV-1 infection as documented by any licensed ELISA test kit within 21 days prior to study entry.
* Age greater than or equal to 18 but less than or equal to 60 years.
* Ability and willingness to give written informed consent.
* Within 30% (+/-) of ideal body weight and total body weight of ≥ 50 kg.
* Hematology, Metabolic Profile, Renal, and Hepatic Function tests all within normal limits.
* Creatine kinase (CK) less than 3 times the upper limit of normal

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Women and men of reproductive potential who are actively engaging in sexual activity or assisted reproductive technology with the intent of pregnancy.
* Allergy/sensitivity to raltegravir.
* Allergy/sensitivity to antacids.
* Active drug or alcohol abuse or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements. While on study, subjects will be instructed not to consume alcohol for 48 hours prior the screening visit, and for the 24 hours preceding the intensive pharmacokinetic (PK) study visits and for 24 hours following the completion of the study visits.
* Any medical condition that, in the opinion of the investigator, would interfere with the subject's ability to participate in this protocol.
* Participation in any investigational drug studies within 30 days prior to study entry.
* History of or active cardiovascular, renal, hematologic, hepatic, neurologic, gastrointestinal, psychiatric, endocrine, or immunologic disease(s). This is inclusive of chronic illnesses such as hypertension, coronary artery disease, arthritis, diabetes, any chronic gastrointestinal conditions that might interfere with drug absorption.
* Use of investigational, prescription, and over-the-counter medications within 14 days of study entry with the following exceptions: aspirin, acetaminophen, ibuprofen, and oral contraceptives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Raltegravir AUC with and without an antacid | 0-48 hours

SECONDARY OUTCOMES:
Raltegravir Cmax with and without an antacid | 0-48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Kiser, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States